CLINICAL TRIAL: NCT00345826
Title: Long-Term Safety and Efficacy of Dasatinib (BMS-354825) in Subjects Who Experienced Clinical Benefit on Protocol CA 180-002
Brief Title: Dasatinib in Treating Patients With Chronic Myelogenous Leukemia or Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000480396; UCLA-0509010-01; BMS-CA180039
Record Dates: First submitted 2006-06-28; First posted 2006-06-29 (Estimated); Last update posted 2013-01-08 (Estimated); Status verified 2013-01

CONDITIONS: Leukemia
Keywords: accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; chronic phase chronic myelogenous leukemia; relapsing chronic myelogenous leukemia; recurrent adult acute lymphoblastic leukemia; chronic myelogenous leukemia, BCR-ABL1 positive
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Leukemia, Myeloid, Chronic-Phase; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dasatinib (Experimental)
  Interventions: Drug: dasatinib

INTERVENTIONS:
Drug: dasatinib

SUMMARY:
RATIONALE: Dasatinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This phase I trial is studying the side effects of dasatinib in treating patients with chronic myelogenous leukemia or acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the long-term safety and tolerability of dasatinib in patients with Philadelphia chromosome-positive chronic myelogenous leukemia or acute lymphoblastic leukemia resistant or intolerant to imatinib mesylate.

Secondary

* Describe any hematologic or cytogenetic response in patients treated with this drug.
* Determine the duration of hematologic and cytogenetic response in patients using this drug during trial UCLA-0303035.
* Determine the progression-free survival and overall survival of patients treated with this drug.

OUTLINE: This is an open-label, roll-over study of protocol UCLA-0303035.

Patients receive oral dasatinib once or twice daily for 5, 6, or 7 days. Treatment repeats every 7 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically for 5 years.

PROJECTED ACCRUAL: A total of 54 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of one of the following hematologic malignancies:

  * Chronic phase chronic myelogenous leukemia (CML)

    * In complete hematologic response after treatment on protocol UCLA-0303035, as indicated by the following criteria:

      * WBC ≤ upper limit of normal (ULN)
      * Platelet count < 450,000/mm^3
      * No blasts or promyelocytes in peripheral blood
      * Less than 5% myelocytes plus metamyelocytes in peripheral blood
      * Peripheral blood basophils ≤ ULN
      * No extramedullary involvement (including no hepatomegaly or splenomegaly)
      * Response lasting ≥ 4 weeks after first documentation
  * Accelerated or blastic phase CML or acute lymphoblastic leukemia

    * In major hematologic response* after treatment on protocol UCLA-0303035, defined as 1 of the following:

      * In complete hematologic response*, as indicated by the following criteria:

        * WBC ≤ ULN
        * Absolute neutrophil count ≥ 1,000/mm^3
        * Platelet count ≥ 100,000/mm^3
        * No blasts or promyelocytes in peripheral blood
        * Bone marrow blasts ≤ 5%
        * Less than 5% myelocytes plus metamyelocytes in peripheral blood
        * Peripheral blood basophils ≤ ULN
        * No extramedullary involvement (including no hepatomegaly or splenomegaly)
      * No evidence of leukemia, as indicated by the following criteria:

        * WBC ≤ ULN
        * No blasts or promyelocytes in the peripheral blood
        * Bone marrow blasts ≤ 5%
        * Less than 5% myelocytes plus metamyelocytes in peripheral blood
        * Peripheral blood basophils ≤ ULN
        * No extramedullary involvement (including no hepatomegaly or splenomegaly)
        * Absolute neutrophil count ≥ 500/mm^3 and < 1,000/mm^3 AND platelet count ≥ 20,000/mm^3 and < 100,000/mm^3
    * In minor hematologic response* after treatment on protocol UCLA-0303035, as indicated by the following criteria:

      * Less than 15% in bone marrow and < 15% in peripheral blood
      * Less than 30% blasts plus promyelocytes in bone marrow and < 30% blasts plus promyelocytes in peripheral blood
      * Less than 20% basophils in peripheral blood
      * No extramedullary disease other than spleen and liver NOTE: *Response confirmed after ≥ 4 weeks allowed provided there is no concurrent anagrelide or hydroxyurea during this time
* Philadelphia chromosome-positive (Ph+) disease
* Resistant or intolerant to prior imatinib mesylate
* Received and benefitted from ≥ 3 months of prior therapy with dasatinib on protocol UCLA-0303035

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 12 weeks after completion of study treatment
* No serious uncontrolled medical disorder
* No active infection that would preclude study participation
* No uncontrolled angina within the past 3 months
* No diagnosed or suspected congenital long QT syndrome
* No history of clinically significant ventricular arrhythmias (e.g., ventricular tachycardia, ventricular fibrillation, or torsades de pointes)
* QTc ≤ 450 msec on electrocardiogram
* No uncontrolled hypertension
* No dementia or altered mental status the would prohibit the understanding or rendering of informed consent
* No history of the following significant bleeding disorders unrelated to CML:

  * Diagnosed congenital bleeding disorders (e.g., von Willebrand's disease)
  * Diagnosed acquired bleeding disorder in the past year (e.g., acquired antifactor VIII antibodies)
* Not involuntarily incarcerated for either psychiatric or physical (e.g., infectious disease) illness
* No patients who are imprisoned
* No clinical adverse event, laboratory abnormality, or intercurrent illness that may preclude study treatment, in the opinion of the investigator
* Bilirubin < 1.5 mg/dL
* ALT and AST < 2 times upper limit of normal (ULN)
* Creatinine < 1.5 times ULN

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No concurrent use of the following drugs that may confer risk of torsades de pointes:

  * Quinidine
  * Procainamide
  * Disopyramide
  * Amiodarone
  * Sotalol
  * Ibutilide
  * Dofetilide
  * Erythromycin
  * Clarithromycin
  * Chlorpromazine
  * Haloperidol
  * Mesoridazine
  * Thioridazine
  * Pimozide
  * Cisapride
  * Bepridil
  * Droperidol
  * Methadone
  * Arsenic
  * Chloroquine
  * Domperidone
  * Halofantrine
  * Levomethadyl
  * Pentamidine
  * Sparfloxacin
  * Lidoflazine
* No other concurrent treatment for CML except for hydroxyurea for a 2-week duration
* No concurrent medications that inhibit platelet function (e.g., aspirin, dipyridamole, epoprostenol, eptifibatide, clopidogrel, cilostazol, abciximab, ticlopidine, or any nonsteroidal anti-inflammatory drug)* except for hydroxyurea or anagrelide
* No concurrent anticoagulants (e.g., warfarin or heparin/low molecular weight heparin [e.g., danaparoid, dalteparin, tinzaparin, or enoxaparin]) except as prophylaxis for catheter thrombosis and/or heparin flushes for IV lines* NOTE: *Allowed if received previously on UCLA-0303035

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2005-11; Primary Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Long term safety and tolerability | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Charles Sawyers, MD, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California, United States

REFERENCES:
- [Result] Talpaz M, Shah NP, Kantarjian H, Donato N, Nicoll J, Paquette R, Cortes J, O'Brien S, Nicaise C, Bleickardt E, Blackwood-Chirchir MA, Iyer V, Chen TT, Huang F, Decillis AP, Sawyers CL. Dasatinib in imatinib-resistant Philadelphia chromosome-positive leukemias. N Engl J Med. 2006 Jun 15;354(24):2531-41. doi: 10.1056/NEJMoa055229. PMID 16775234